CLINICAL TRIAL: NCT02300506
Title: Post-Marketing Surveillance of Long-Term Observation of Gliadel Wafer-Investigation of Vital Prognosis in Patients With High Grade Glioma
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: GLI02T
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2017-08

CONDITIONS: Malignant Glioma
Keywords: Malignant Glioma; Glioblastoma multiforme
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with diagnosed malignant glioma treated by surgery, implanted Gliadel wafers 7.7mg, and enrolled in study GLI01S.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The objective of this study is to determine the survival status of patients enrolled in study GLI01S (all-case observational study).

ELIGIBILITY:
Inclusion criteria:

* Malignant Glioma, patients enrolled in study GLI01S.

Exclusion criteria:

* Corresponding to contraindication of Gliadel.
* Not applicable to indications of Gliadel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosed malignant glioma treated by surgery
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2016-07-10 (Actual)

PRIMARY OUTCOMES:
Survival rate | Up to 3 years
  Survival rate of subjects measured up to 3 year after implantation

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

REFERENCES:
- [Derived] Iuchi T, Inoue A, Hirose Y, Morioka M, Horiguchi K, Natsume A, Arakawa Y, Iwasaki K, Fujiki M, Kumabe T, Sakata Y. Long-term effectiveness of Gliadel implant for malignant glioma and prognostic factors for survival: 3-year results of a postmarketing surveillance in Japan. Neurooncol Adv. 2022 Jan 12;4(1):vdab189. doi: 10.1093/noajnl/vdab189. eCollection 2022 Jan-Dec. PMID 35118382